CLINICAL TRIAL: NCT01552499
Title: A Prospective, Randomized, Comparative Parallel Study of Amniotic Membrane Wound Graft In the Management of Diabetic Foot Ulcers
Brief Title: Comparative Study of Amniotic Membrane Wound Graft In the Management of Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MiMedx Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: EFDFU001
Record Dates: First submitted 2012-03-06; First posted 2012-03-13 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

ARMS (2):
- Control (Other)
  Interventions: Other: Standard of care
- Treatment (Experimental)
  Interventions: Other: Standard of care; Other: Applications of EpiFix

INTERVENTIONS:
Other: Standard of care
Other: Applications of EpiFix
  Arms: Treatment

SUMMARY:
The purpose of this study is to determine whether the EpiFix human amniotic membrane is effective in the treatment of diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18 or older
* Informed consent must be obtained
* Patient's ulcer must be diabetic in origin and larger than 1cm2. Debridement will be done prior to randomization. Subject's informed consent for participating in this study, must be obtained prior to proceeding with sharp debridement.
* Patients with Type 1 or Type 2 diabetes (criteria for the diagnosis of diabetes mellitus per ADA).
* Ulcer must be present for a minimum of four weeks direction, with documented failure of prior treatment to heal the wound.
* Patient's ulcer must exhibit no clinical signs of infection.
* Patient is of legal consenting age.
* Patient is willing to provide informed consent and is willing to participate in all procedures and follow up evaluations necessary to complete the study.
* Serum Creatine less then 3.0mg/dl
* HbA1c less than 12%
* Patient has adequate circulation to the affected extremity, as demonstrated by one of the following within the past 60 days:

  * Dorsum transcutaneous oxygen test (TcPO2) with results ≥30mmHg, OR
  * ABIs with results of ≥0.7 and ≤1.2, OR
  * Doppler arterial waveforms, which are triphasic or biphasic at the ankle of affected leg

Exclusion Criteria:

* Patients presenting with an ulcer probing to bone (UT Grade IIIA-D). A positive probe-to-bone will be confirmed when bone or joint can be felt with a sterile, ophthalmological probe.
* Patients whose index diabetic foot ulcers are greater than 25cm2.
* Patients considered not in reasonable metabolic control, confirmed by an HbA1c greater than 12% within previous 90 days,
* Patients whose serum creatinine levels are 3.0mg/dl or greater.
* Patients with a known history of poor compliance with medical treatments.
* Patients who have been previously randomized into this study, or are presently participating in another clinical trial.
* Patients who are currently receiving radiation therapy or chemotherapy.
* Patients with known or suspected local skin malignancy to the index diabetic ulcer.
* Patients on anticoagulant medication will as in any surgical procedure, be monitored according to the protocols employed at the enrolling center.
* Patients diagnosed with autoimmune connective tissues diseases.
* Non-revascularizable surgical sites.
* Active infection at site.
* Any pathology that would limit the blood supply and compromise healing.
* Patients that have received a biomedical or topical growth factor for their wound within the previous 30 days.
* Patient who are pregnant or breast feeding.
* Patient who are taking medications that are considered immune system modulator which could affect graft incorporation.
* Allergy to Gentamycin or Streptomycin.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
The proportion of completely healed ulcers in patients treated with amniotic membrane vs. standard of care | 12 week

SECONDARY OUTCOMES:
Percent change in wound area | 4 week
Mean time to complete healing | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Charles M. Zelen, DPM, Principal Investigator — Professional Education and Research Institute
Locations (1):
- Professional Education and Research Institute, Roanoke, Virginia, United States